CLINICAL TRIAL: NCT00873964
Title: Metabolic Syndrome in an Elderly Population is More Linked to Insulin Resistance Than to Obesity
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Terre Williams, Research assistant, Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Other Study IDs: HM11534
Record Dates: First submitted 2009-04-01; First posted 2009-04-02 (Estimated); Last update posted 2012-04-30 (Estimated); Status verified 2012-04

CONDITIONS: Metabolic Syndrome in the Elderly
Keywords: Metabolic Syndrome; Obesity; Elderly; Insulin Resistance
MeSH Terms: conditions — Metabolic Syndrome; Obesity; Insulin Resistance

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum collected.
Oversight: Data Monitoring Committee: No

SUMMARY:
In the United States cardiovascular disease (CVD) accounts for 1 in every 2.8 deaths and is the leading cause of death among men and women 65 years or older (1). Studies have shown that the risk for cardiovascular disease is higher in individuals with the Metabolic Syndrome (2). Metabolic Syndrome (MBS) is defined by the Adult Treatment Panel III (ATP III) guidelines as a group of risk factors that includes 3 or more of the following: abdominal obesity, hypertriglyceridemia, low high-density lipoprotein (HDL) cholesterol, high blood pressure, and high fasting glucose (3). These factors place individuals at increased risk for the development of both cardiovascular disease (CVD) and diabetes mellitus (3). It is commonly held that insulin resistance is the driving force for the development of the MBS.

Although there is a significant increase in incidence of MBS in the elderly, there are few studies that specifically examined MBS in that population. The prevailing opinion is that the strikingly high prevalence of the MBS in the elderly is due to concurrent obesity - i.e., the population gains weight as it ages, and development of the MBS accompanies the weight gain.

However, while it is true that becoming obese may decrease insulin sensitivity, it has also been demonstrated that not all obese individuals are insulin resistant. Some studies suggest that up to 40% of obese individuals demonstrate normal insulin sensitivity (4). In addition, it is notable that the rate of increasing MBS in the population exceeds that of the rate of increasing BMI, suggesting that, while BMI may be a modulating factor, another factor independent of obesity also contributes to the development of MBS in the elderly.

It is the investigators hypothesize that the MBS in the obese elderly population is primarily linked to insulin resistance and not to obesity per se. The investigators propose to test this hypothesis by assessing MBS and insulin resistance in a population of obese elderly men and women and then determining whether or not the MBS tracks with insulin resistance.

ELIGIBILITY:
Inclusion Criteria:

* Approximately 156 obese (BMI 30-34 kg/m2) non-diabetic men and women between the ages of 60-80 years of age will be eligible to enroll in the study if they meet the following inclusion criteria:

  * BMI 30-34 kg/m2
  * Ability and willingness to provide signed, witnessed informed consent.

Exclusion Criteria:

* Diabetes mellitus. WHO diagnostic criteria for diabetes mellitus is fasting plasma glucose > 7.0 mmol/l (126 mg/dl) or 2-h plasma glucose > 11.1 mmol/l (200mg/dl).
* Subjects in this group experience increased premature mortality and increased risk of microvascular and cardiovascular complications (25).
* Subjects with clinically apparent cardiovascular disease including prior history of cardiac angina, MI, interventional percutaneous procedures, coronary artery bypass graft, congestive heart disease, cerebral vascular accident, peripheral vascular disease, and pulmonary embolus.
* Subjects with serum creatinine greater than 3.
* Subjects with moderate or severe COPD or on home oxygen.
* Subjects with serum total bilirubin greater than 4.
* Subjects with concurrent infectious disease.
* Subjects with malignancy (except for prostate ca, or basal cell carcinoma of the skin) diagnosed within the last year, or on concurrent chemotherapy.
* Subjects receiving androgen or anti-androgen therapy.
* Hormone replacement therapy.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Approximately 156 obese (BMI 30-34 kg/m2), non-diabetic men and women between the ages of 60-80 years of age will be eligible to enroll in the study if they meet the following inclusion criteria: (1) BMI 30-34 kg/m2. (2) Ability and willingness to provide signed, witnessed informed consent.
Sampling Method: Probability Sample
Enrollment: 156 (Estimated)
Dates: Start 2009-03; Primary Completion 2013-04 (Estimated); Study Completion 2013-07 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- McGuire VAMC, Richmond, Virginia, United States